CLINICAL TRIAL: NCT03170089
Title: Effect of Oral Health Educational Program on Awareness and Oral Health Status of Children With Insulin Dependent Diabetes Mellitus: A Randomized Clinical Trial
Brief Title: Oral Health Awareness and Oral Hygiene in Insulin Dependent Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samar Ali Zein El Abdeen Haikal, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S.Haikal
Record Dates: First submitted 2017-05-17; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Health Attitude; Diabetes type1
Keywords: oral-health-awareness, Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Professional tooth cleaning (scaling) Oral Health educational program
  Interventions: Behavioral: Oral Health Educational Program
- Control (No Intervention): NO program or scaling done

INTERVENTIONS:
Behavioral: Oral Health Educational Program — Oral Hygiene methods learned
  Arms: Intervention

SUMMARY:
This study is designed to evaluate the effect of oral health educational program on the awareness and oral health status of children with Insulin Dependent Diabetes Mellitus.

DETAILED DESCRIPTION:
First visit: (baseline)

1. Awareness questionnaire is given to parent or caregiver to fill.
2. Child information will be recorded in the diagnosis chart of Pediatric Dentistry and Public Health Department
3. Intra-oral and extra-oral examination to all children included and recording Oral Hygiene Index simplified.
4. Intervention group will receive:

   * Supra-gingival scaling
   * Oral Health Educational Program through life demonstration of tooth brushing on a model, power point presentation and a poster.
   * Package containing tooth brush, tooth paste, poster and follow-up chart.

Second and third visits: (every month)

1. Oral hygiene index simplified will be recorded for both groups.
2. Follow-up chart is collected from intervention group.

Forth visit: (final visit)

1. Awareness questionnaire is given for parents of both groups.
2. Oral Hygiene Index simplified is recorded for both groups.
3. Follow up charts is collected from intervention
4. Control group will receive the same program after collection all data.

Number of visits & follow up period:

* Four visits, time interval between each visit is one month and the follow up period is three months

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 6-8 years old.
2. Cooperative children.
3. Both genders.
4. Insulin Dependent Diabetes Mellitus children

Exclusion Criteria:

1. Children with any other medical condition.
2. Children undergoing orthodontic treatment.
3. Parents unable to give informed consent

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2017-06-30 (Estimated); Primary Completion 2017-10-30 (Estimated); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
Patient awareness | Baseline
  Questionnaire about oral health

SECONDARY OUTCOMES:
Oral hygiene | 3 months
  Oral Hygiene Index- Simplified

CONTACTS AND LOCATIONS:
Overall Officials: Fatma El-Shehaby, Professor, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: No